CLINICAL TRIAL: NCT01652287
Title: Yogurt Beverages as a Vehicle to Deliver High Dose Probiotics
Brief Title: Safety of BB-12 Supplemented Strawberry Yogurt For Healthy Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Penn State University (Other)
Responsible Party: Principal Investigator, Daniel Merenstein, Principal Investigator, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 3U01AT003600-02S1 (NIH)
Record Dates: First submitted 2012-07-05; First posted 2012-07-30 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-02

CONDITIONS: Children

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BB-12 supplemented yogurt (Active Comparator): Probiotic, Bifidobacterium animalis subsp. lactis (B. lactis) strain BB-12 (BB-12), supplemented strawberry yogurt, 4 ounces taken orally for 10 days
  Interventions: Drug: BB-12 supplemented strawberry yogurt
- Strawberry flavored yogurt (Placebo Comparator): Placebo, strawberry yogurt, 4 ounces taken orally for 10 days
  Interventions: Other: Strawberry flavored yogurt

INTERVENTIONS:
Drug: BB-12 supplemented strawberry yogurt — Bifidobacterium animalis subsp. lactis (B. lactis) strain BB-12 (BB-12) probiotic supplemented yogurt, 4 ounces taken orally for 10 days
  Arms: BB-12 supplemented yogurt
Other: Strawberry flavored yogurt — Placebo, strawberry yogurt, 4 ounces taken orally for 10 days
  Arms: Strawberry flavored yogurt

SUMMARY:
The investigators believe a readily available drink containing a high dose of probiotics has the potential to improve compliance through many of these mechanisms. This product also has the potential to positively impact the health of children and adults around the world, as yogurt will likely be more appealing to both children and their parents for long term consumption than pharmaceutical-like preparations. In addition to the benefits associated with the consumption of probiotics, there is an increased health benefit from consuming yogurt, a nutrient dense food.

More specifically, the rationale for this Phase I study is to determine safety of this yogurt drink and comply with FDA recommendations pertaining to an Investigational New Drug application. The investigators hypothesize that BB-12 is safe in generally healthy children ages 1-5 years.

DETAILED DESCRIPTION:
Probiotics are live microorganisms that, when administered in sufficient amounts, may improve health. A common use for probiotics is in addressing gastrointestinal issues, such as antibiotic-associated diarrhea (AAD). As an alternative to supplements, probiotics are also included as ingredients in fermented dairy products to produce functional foods, which are foods providing health benefits beyond their nutritional value. Yogurt, for example, is a fermented milk product often considered a functional food. One of the most commonly used probiotics is Bifidobacterium animalis ssp. lactis (BB-12).

Our Primary Aim in Years 1-2 is to conduct a pediatric randomized controlled study to establish the safety of BB-12 fortified yogurt in children. Our Secondary Aims are to examine the fecal microbiota of children prior to, during and following consumption of probiotics. This study will evaluate whether a well-defined, probiotic-containing yogurt can safely be used as an effective delivery vehicle for probiotics. This study is important to help advance probiotic research forward in a systematic, well-accepted manner. Our long-term goal is to create yogurt with sufficient probiotic dosages to positively impact many different aspects of childhood and adult health.

ELIGIBILITY:
Inclusion criteria for parents/caregivers are:

1. Ability to read, speak and write English or Spanish
2. Access to a refrigerator for proper storage of drink
3. Telephone access

Inclusion criteria for children are:

1. Are between the ages of 1 and 5 years

Exclusion Criteria:

1. Developmental delays
2. Any chronic condition, such as diabetes or asthma, that requires medication
3. Prematurity, birth weight < 2,500 grams
4. Congenital anomalies
5. Failure to thrive
6. Allergy to strawberry
7. Active diarrhea (defined as three or more loose stools for two consecutive days)
8. Any other medicines used except anti-pyretic medicines (to reduce fever) [excluding as needed medications]
9. Parental belief of lactose intolerance
10. History of heart disease, including valvulopathies or cardiac surgery, any implantable device or prosthetic
11. History of gastrointestinal surgery or disease
12. Milk-protein allergy
13. Allergy to any component of the product or the yogurt vehicle
14. During the baseline physical exam, have an oxygen saturation rate <96% and respiratory and pulse rate outside the normal range per their age.

Parents/caregivers will also be asked to refrain from giving their child any probiotic foods or supplements during the entire 2 weeks of the active intervention period, and 2 weeks before day 1 of starting the yogurt. Parents will be supplied with a list of products to avoid.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Merenstein, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Department of Family Medicine, Research Division, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Tan TP, Ba Z, Sanders ME, D'Amico FJ, Roberts RF, Smith KH, Merenstein DJ. Safety of Bifidobacterium animalis Subsp. Lactis (B. lactis) Strain BB-12-Supplemented Yogurt in Healthy Children. J Pediatr Gastroenterol Nutr. 2017 Feb;64(2):302-309. doi: 10.1097/MPG.0000000000001272. PMID 28114246

RESULTS

PARTICIPANT FLOW:
Groups:
- BB-12: Bifidobacterium animalis subsp. lactis (B. lactis) strain BB-12®-supplemented yogurt
- Control: yogurt cultured with starter YF-L702
Period: Overall Study
Arm/Group | BB-12 | Control
Started | 31 | 31
Completed | 29 (• Did not receive allocated intervention (withdrew consent) (n=2)) | 31
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- BB-12®: Bifidobacterium animalis subsp. lactis (B. lactis) strain BB-12®-supplemented yogurt
- Total: Total of all reporting groups
Arm/Group | BB-12® | Control | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29 | 31 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 31
  Male | 16 | 13 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 26 | 26 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 21 | 17 | 38
  More than one race | 1 | 6 | 7
  Unknown or Not Reported | 0 | 0 | 0
Child Attends Daycare [Count of Participants; unit: Participants]
  Yes | 20 | 17 | 37
  No | 9 | 14 | 23
Parent's Marital Status [Count of Participants; unit: Participants]
  Married/Living with partner | 26 | 28 | 54
  Single | 3 | 1 | 4
  Divorced | 0 | 2 | 2
Total Household Income [Count of Participants; unit: Participants]
  $15,000-$30,000 | 2 | 1 | 3
  $30,001-$75,000 | 6 | 10 | 16
  $75,001-$100,000 | 6 | 6 | 12
  $100,001-$150,000 | 8 | 8 | 16
  >$150,000 | 6 | 6 | 12
  No response | 1 | 0 | 1
Smoker in Household-Yes [Count of Participants; unit: Participants] | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: The primary outcome is to assess the safety of BB-12® yogurt when consumed by generally healthy children. To achieve this aim, data on adverse events will be collected from diaries; calls to the 24-hour advice line; and research assistant phone calls on days 6, 11, 15 and 180, ±2 days. All adverse events will be tabulated by type and charted over time.
Time Frame: Days 0-180
Measure: Number; unit: Number of AE reported
Arm/Group | BB-12® | Control
Number analyzed (Participants) | 29 | 31
Number of AE reported
  During intervention (day 0-10) | 61 | 35
  Post-intervention (day 11-180) | 52 | 38

2. Secondary Outcome: Overall Composition of the Gut Microbiota
Description: Relative abundance of operational taxonomic units (OTU) classified at the phylum level
Time Frame: 90 days
Measure: Number; unit: relative abundance (%)
Arm/Group | BB-12 | Control
Number analyzed (Participants) | 29 | 31
relative abundance (%)
  Firmicutes | 71.7 | 74.1
  Bacteroidetes | 14.7 | 11.6
  Actinobacteria | 11.1 | 11.9
  Proteobacteria | 1.6 | 1.4
  Verrucomicrobia | 0.7 | 1.0

ADVERSE EVENTS:
Arm/Group | BB-12® | Control
Serious Adverse Events (participants affected / at risk) | 3/29 | 0/31
Other Adverse Events (participants affected / at risk) | 22/29 | 22/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BB-12® (N=29) | Control (N=31)
Fever (General disorders) | 1 (1) | 0 (0)
bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BB-12® (N=29) | Control (N=31)
Runny nose (General disorders) | 17 (21) | 10 (12)
Other (General disorders) | 5 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes